CLINICAL TRIAL: NCT06814288
Title: The Effectiveness of Intralesional Botulinum Toxin A and Triamcinolone Acetonide Injections in Keloid Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DV-202501.01
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Keloid Scars
Keywords: Keloid; Botulinum Toxin A; Triamcinolone Acetonide; Intralesional Injection
MeSH Terms: conditions — Keloid | interventions — Botulinum Toxins, Type A; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin A (Experimental): Twenty keloid patients will be injected botulinum toxin A intralesional every 4 weeks.
  Interventions: Drug: Botulinum toxin A
- Triamcinolone Acetonide (Active Comparator): Twenty keloid patients will be injected triamcinolone acetonide intralesional every 4 weeks.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Botulinum toxin A — Twenty keloid patients will be injected botulinum toxin A intralesional every 4 weeks.
  Arms: Botulinum Toxin A
Drug: Triamcinolone Acetonide — Twenty keloid patients will be injected triamcinolone acetonide intralesional every 4 weeks.
  Arms: Triamcinolone Acetonide

SUMMARY:
Keloids are benign fibrous tissue overgrowths that extend beyond the boundaries of the original wound and tend to recur after therapy. The exact pathogenesis of keloids is not fully understood; however, the role of TGF-β leads to an imbalance in collagen synthesis and degradation, while VEGF increases vascularity. Enhanced vascularity contributes to increased fibroblast activity. Angiogenesis is heightened in wounds subjected to high tension. Active keloids are characterized by low vascular velocity, low elasticity, and varied echogenicity depending on the filling tissue, as observed on ultrasonographic examination. Intralesional TA injections at 40 mg/ml are an available option for keloids, but this therapy is associated with various side effects. Intralesional TB-A injections at 5 U/cm³ have been reported to demonstrate good efficacy, safety, tolerable side effects, and high patient satisfaction for keloid management. Therefore, it is necessary to conduct a study comparing the effectiveness of intralesional TB-A injections at 5 U/cm³ with intralesional TA injections at 40 mg/ml in keloid patients. Scar assessment can generally be conducted objectively using various tools or subjectively through different measurement scales. The Japan Scar Workshop (JSW) developed a measurement scale known as the JSW scar scale (JSS).

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of intralesional TB-A injections at 5 U/cm³ compared to intralesional TA injections at 40 mg/ml in keloid patients in Indonesia, assessed using the Japan Scar Scale (JSS) and measurements of lesion volume, vascularization degree, vascular velocity, elasticity, and echogenicity through high-resolution ultrasonography. Such research has not been conducted before.

The study design is an experimental single-blind randomized trial with a pretest-posttest design. Participants include keloid patients seeking treatment at the Tumor and Dermatologic Surgery Clinic, Department of Dermatology and Venereology, RSHS Bandung, who meet the inclusion and exclusion criteria. Lesions and treatments are randomized by the researchers, and the selected treatment is then administered to the keloid lesions. Observations are repeated to evaluate the effectiveness of the therapy using JSS and high-resolution ultrasonography.

During patient visits, the following procedures are conducted:

History Taking and Physical Examination Patients undergo anamnesis and a thorough physical examination.

Baseline Keloid Lesion Measurement Initial lesion measurements are performed using a caliper to establish baseline data before therapy.

Elasticity Measurement Baseline lesion elasticity is measured using the Cutometer MPA 580 at the midpoint of each lesion. Skin erythema is assessed using the CM-700d Spectrophotometer.

High-Resolution Ultrasonography Assessment

A radiology specialist performs the ultrasonography using a Phillips EPIQ Elite® high-resolution ultrasound device with a linear transducer at 22 MHz. The machine's automatic settings for observing superficial structures are applied uniformly across cases.

Patients are positioned upright or lying down, depending on lesion location. The transducer is placed perpendicularly to the keloid lesion in both transverse and longitudinal orientations without applying pressure.

Measurements include lesion volume, vascularization degree, vascular velocity, elasticity, and echogenicity type.

Documentation involves recording data and capturing images on the ultrasound machine.

Photographic Documentation Lesions are photographed from the top and side for documentation.

Randomization and Group Assignment

Lesions are randomly assigned to one of two therapy groups:

Group I: Intralesional Botulinum Toxin A injection at 5 U/cm³. Group II: Intralesional Triamcinolone Acetonide injection at 40 mg/ml. These detailed procedures ensure a comprehensive evaluation of the comparative efficacy of the two treatments in managing keloid lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients aged ≥ 18 years.
2. Patients clinically diagnosed with keloids.
3. Patients with at least two keloid lesions located on different sides but in similar anatomical regions.
4. Keloid lesion size is limited to ≤ 5 cm².
5. All keloid patients who will not undergo other keloid treatments (surgical excision, chemotherapy injections, laser therapy, radiation therapy, cryotherapy, or pressure therapy) during the study and observation period.
6. All keloid patients who have not undergone any keloid treatment in the past two months.

Exclusion Criteria:

1. Pregnant and breastfeeding women.
2. Patients currently using hormonal contraceptives.
3. Patients undergoing long-term systemic corticosteroid therapy.
4. History of hypersensitivity to botulinum toxin.
5. Use of or exposure to aminoglycosides, lincosamides, polymyxins, quinine, magnesium sulfate, anticholinesterases, succinylcholine, or other serotypes of botulinum toxin.
6. Presence of motor peripheral neuropathy (e.g., amyotrophic lateral sclerosis or motor neuropathy), neuromuscular junction disorders (e.g., myasthenia gravis or Lambert-Eaton syndrome), diabetes mellitus, or uncontrolled cardiovascular disorders.
7. Infection at the injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Japan Scar Workshop Scar Scale (JSS) | 12 weeks
  Evaluation for Groups I and II is conducted every four weeks, specifically in the 4th, 8th, and 12th weeks. At each visit, assessments of JSS for evaluation consists of six items: (1) Induration, (2) Elevation, (3) Redness of the scar, (4) Erythema around the scar, (5) Spontaneous and pressing pain, and (6) Itch. Each item has four intensity categories, namely, None, Weak, Mild, and Strong. These categories are weighted 0, 1, 2, and 3, respectively. There are sample images of each category in each item that helps the user judge the items. The minimum and maximum total points in the evaluation table are thus 0 and 18, respectively. When the symptoms improve, the total score decreases.
Lesion volume by ultrasonography | 12 weeks
  Lesion volume in mililiters (ml) are measured by high-resolution ultrasonography on the initial visit (before therapy) and week-12 (after therapy)
Elasticity | 12 weeks
  Elasticity ratio between keloid lesion and normal skin are measured by cutometer and high-resolution ultrasonography on the initial visit (before therapy) and week-12 (after therapy)
Echogenicity on ultrasonography | 12 weeks
  Echogenicity of keloid lesion are measured by high-resolution ultrasonography on the initial visit (before therapy) and week-12 (after therapy)
Degree of Vascularity on ultrasonography | 12 weeks
  Degree of Vascularity of keloid lesion are measured by high-resolution ultrasonography on the initial visit (before therapy) and week-12 (after therapy)

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) after every injection session | 12 weeks
  Evaluation for Groups I and II is conducted every four weeks, specifically in the 4th, 8th, and 12th weeks. At each visit, assessments of VAS for therapy evaluation
Adverse Effects | 12 weeks
  Evaluation of any adverse effects for Groups I and II is conducted every four weeks, specifically in the 4th, 8th, and 12th weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva K sutedja, M.D., Principal Investigator — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia